CLINICAL TRIAL: NCT03223350
Title: Topical Capsaicin Cream for Treatment of Suspected Cyclical Vomiting Syndromes
Brief Title: Topical Capsaicin for Cyclical Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Joseph Miller, MD, Senior Staff, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10658
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Cyclical Vomiting
MeSH Terms: conditions — Familial cyclic vomiting syndrome | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical appearing placebo cream used for control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Capsaicin (Experimental): 0.1% capsaicin cream, one application
  Interventions: Drug: Capsaicin 0.1% Cream
- Placebo (Placebo Comparator): Topical cream with no active drug
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Capsaicin 0.1% Cream — Topical application
  Arms: Capsaicin
Drug: Placebos — placebo cream
  Arms: Placebo

SUMMARY:
This is a phase 2 randomized controlled trial testing the effect of topical capsaicin for the relieve of nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* suspected cyclical vomiting syndrome / cannabinoid hyperemesis
* active severe nausea or vomiting in the emergency department

Exclusion Criteria:

* pregnant women, children < 18 years, no prior history of similar symptoms, suspected surgical or infectious cause of symptoms, suspected hepatitis or pancreatitis, allergy to capsaicin or hot peppers, chronic use of prescription antiemetic in prior 24 hours, abdominal pain alone (without nausea or vomiting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Miller, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capsaicin | Placebo
Started | 17 | 13
Completed | 17 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capsaicin | Placebo | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (15.3) | 27.5 (5.2) | 32.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 1 | 1 | 2
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30
Nausea on visual analog scale [Mean (Standard Deviation); unit: mm] — Minimum measurement 0, maximum 100. Higher score indicates more severe nausea.
  mm | 60 (29) | 85 (20) | 71 (28)

OUTCOME MEASURES:

1. Primary Outcome: Nausea Visual Analog Scale
Description: Nausea visual analog scale, ranging from 0-100 mm, high measurement indicates worse nausea
Time Frame: 30 minutes
Population: Patients identified with cannabinoid hyperemesis
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Capsaicin | Placebo
Number analyzed (Participants) | 17 | 13
mm | 41 [28 to 54] | 61 [41 to 81]

ADVERSE EVENTS:
Time Frame: 4 hours
Arm/Group | Capsaicin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 1/17 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capsaicin (N=17) | Placebo (N=13)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03223350/Prot_002.pdf
  • Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT03223350/SAP_003.pdf